CLINICAL TRIAL: NCT06645678
Title: Phase I/II Study of Mezigdomide and Elranatamab for Relapsed/Refractory Multiple Myeloma Patients
Brief Title: Mezigdomide and Elranatamab for Relapsed and/or Refractory Multiple Myeloma
Acronym: MELT-MM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: YOUNGIL KOH (Other)
Responsible Party: Sponsor-Investigator, YOUNGIL KOH, Professor, MD PhD, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2410-028-1576
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Relapsed Refractory Multiple Myeloma (RRMM)
Keywords: R/R MM; Elranatamab; Mezigdomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Elranatamab: C0D1 12mg sc, C0D4 32mg sc, C0D8 76mg sc, then 76mg sc weekly C1-C6, then 76mg sc bi-weekly from C7 for those achieving PR or better response, then 76mg sc q 4weeks from C12 for those achieving CR or better response Mezigdomide: per RP2D qd, D1-21, q 4weeks Dexamethasone: with elranatamab up until C6: 20mg/day C1-3 > 10mg/day D4-6 (for those >= 75 years old, with uncontrolled DM, Hx of intolerance, 10mg/day -> 5mg/day)
  28days/cycle, 24 cycles (2 years) fixed duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): Participants will receive elranatamab, mezigdomide and dexamethasone.
  Part 1 (safety cohort): approximately 12 participants to select the optimal RP2D and to assess the safety, tolerability, and preliminary efficacy. Every cycle consists of 28 days.
  Part 2 (expansion cohort): approximately 63 participants will be enrolled. The primary objective of Part 2 is to determine the overall response rate per IMWG criteria at 24 months after enrollment.
  Interventions: Drug: Elranatamab; Drug: Mezigdomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elranatamab — Elranatamab: Participants will receive SC administration of elranatamab QW or Q2W. The initial doses of elranatamab will be 12mg (C0D1), 32mg (C0D4), and 76mg (C0D8) and will serve as the 2 step-up priming regimen (Cycle 0). Then, 76mg weekly C1-C6 > then 76mg bi-weekly from C7 for those achieving PR or better > then 76mg q4weeks from C12 for those achieving CR or better response. If the participant subsequently begins to have an increase of disease burden not yet qualifying as PD according to IMWG criteria, dose intervals will return to weekly dosing.
  premedication for Elranatamab: Acetaminophen 650mg (or paracetamol 500mg), Diphenhydramine 25mg (or equivalent), Dexamethasone 20mg (or equivalent).
  In case of mezigdomide discontinuation due to reasons other than disease progression, elranatamab continuation +/- dexamethasone will be allowed until loss of response. The administration of elranatamab +/- dexamethasone will continue per study protocol schedule.
Drug: Mezigdomide — The first day of study treatment dosing with mezigdomide is considered Day 1 of a cycle. (per recommended phase 2 dose, daily [qd], D1-21, q 4weeks). Capsules of mezigdomide will be taken by mouth with or without food.
  In case of elranatamab discontinuation due to reasons other than disease progression, mezigdomide continuation +/- dexamethasone will be allowed until loss of response. The administration of mezigdomide will continue per study protocol.
Drug: Dexamethasone — Administered at the dose of 20 mg/day from C1-3, then 10mg/day from C4-6 as a premedication for elranatamab.
  (for those >=75 yrs, with uncontrolled diabetes mellitus, history of intolerance: 10mg/day -> 5mg/day)

SUMMARY:
The goal of this clinical trial is to find out how well a combination of two medicines (mezigdomide and elranatamab) works in treating patients with refractory/relapsed multiple myeloma.

DETAILED DESCRIPTION:
This is a phase I/II (2 parts), open-label, single arm, multicenter study to evaluate the efficacy and safety of elranatamab in combination with mezigdomide.

Part 1 (safety cohort): Since the combination of elranatamab with mezigdomide has not previously been evaluated, Part 1 (safety cohort) of the study will be conducted in up to approximately 12 participants to select the optimal RP2D and to assess the safety, tolerability, and preliminary efficacy.

Part 2 (expansion cohort): In Part 2 (expansion cohort), approximately 63 participants will be enrolled. The primary objective of Part 2 is to determine the overall response rate per IMWG criteria at 24 months after enrollment. Participants will receive elranatamab, mezigdomide and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:

  * Subject is ≥ 19 years of age at the time of signing the informed consent form (ICF).

    ② Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
    * Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

      ④ Subject has documented diagnosis of MM and measurable disease, defined as any of the following: A. M-protein ≥ 0.5 g/dL by serum protein electrophoresis (sPEP) or B. M-protein ≥ 200 mg/24-hour urine collection by urine protein electrophoresis (uPEP) or C. For subjects without measurable disease in sPEP or uPEP: serum free light chain (sFLC) levels > 100 mg/L (10 mg/dL) involved light chain and an abnormal kappa/lambda FLC ratio.

      *Patients with measurable disease and extramedullary disease will be allowed to participate if there is a measurable extramedullary lesion. These patients require PET-CT follow-up for response evaluation. Those with extramedullary disease (EMD) only will not be allowed to participate: i.e, Patients with plasmacytoma as the only measurable disease are not eligible. For the definition of EMD, refer to Section 8.1.3.

      ⑤ Subject has received 2 or more prior lines of antimyeloma therapy. (Note: One line can contain several phases [e.g., induction, (with or without) hematopoietic stem cell transplant, (with or without) consolidation, and/or (with or without) maintenance therapy).

      ⑥ Subject must have received at least one proteasome inhibitor and lenalidomide.

      ⑦ Subject achieved minimal response or better to at least 1 prior antimyeloma therapy.
      * Subject must have documented disease progression during or after their last antimyeloma regimen.

        ⑨ Subject has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.

        ⑩ Individual of childbearing potential (IOCBP) must: A. Have two negative pregnancy tests as verified by the Investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. This applies even if the subject practices true abstinence* from heterosexual contact.

B. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, 2 forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting study treatment, during the study treatment (including dose interruptions), and for at least 28 days after the last dose of mezigdomide or 150 days after the last dose of elranatamab, whichever is longer.

Note: A IOCBP (Individual of childbearing potential): an individual who: 1) has achieved menarche (first menstrual cycle) at some point; 2) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral salpingectomy (the surgical removal of the fallopian tubes) or oophorectomy (the surgical removal of both ovaries) or 3) has not been naturally postmenopausal (without an alternative medical cause eg, amenorrhea following cancer therapy does not rule out childbearing potential) for at least 12 consecutive months (ie, has had menses at any time during the preceding 12 consecutive months).

⑪ Male subjects must: A. Practice true abstinence* (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant individual or an individual of childbearing potential while participating in the study, during dose interruptions and for at least 28 days after the last dose of mezigdomide whichever is longer, even if he has undergone a successful vasectomy.

* True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

  * Male subjects must agree to refrain from donating sperm while on study treatment, during dose interruptions and for at least 28 days following last dose of mezigdomide,

    * Females must agree to refrain from donating eggs while on study treatment and for at least 28 days after last dose of mezigdomide.

      * Subjects must agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 28 days following the last dose of mezigdomide.

        * Subjects must agree to refrain from receiving live vaccines while on study treatment, during dose interruptions and for at least 90 days following the last dose of the study treatment.

Exclusion Criteria: The presence of any of the following will exclude a subject from enrollment:

* 1 Subject who has had prior treatment with mezigdomide. 2 Patients with gastrointestinal disease or surgery (eg, gastric bypass surgery) that may significantly alter the absorption of mezigdomide and/or other oral study intervention.

  3 Subject who has had prior treatment with anti-BCMA agents (including CAR T-cell therapy, bispecifics and antibodies).

  4 Subject who has had any investigational agents within 28 days or 5 half-lives (whichever is shorter) of initiating study treatment.

A. Participation in another interventional clinical trial concurrent with this study is not permitted, except for those who have completed treatment with the prior investigational agent(s) and are currently in Long-term Follow up.

5 Subject has received any of the following. A. Plasmapheresis within the last 28 days of initiating study treatment B. Major surgery (as defined by the Investigator) within 28 days of initiating study treatment.

C. Radiation therapy, other than local palliative therapy, for myeloma associated bone lesions within 14 days of initiating study treatment.

D. Use of any systemic antimyeloma drug therapy within 14 days of initiating study treatment.

E. Use of potassium competitive acid blockers (eg. tegoprazan, vonoprazan) within 7 days of initiating study treatment.

6 Subject has previously received allogeneic stem cell transplantation within a year during prior therapy or received autologous stem cell transplantation within 12 weeks of initiating study treatment. Patients who received allogeneic stem cell transplantation should not have evidence of active GVHD.

7 Subject has plasma cell leukemia defined by IMWG definition for primary plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or clinically significant light-chain amyloidosis.

8 Subject with known central nervous system (CNS) involvement with myeloma. 9 Subject has any significant medical condition, including active or uncontrolled infection, presence of laboratory abnormality, or psychiatric illness that places the subject at an unacceptable risk for treatment-related complications, if he/she were to participate in the study.

10 Coronavirus disease 2019 (COVID-19) within 7 days for mild or asymptomatic infections or 14 days for moderate/severe infections prior to initiating study intervention. A longer duration may be needed based on the investigator's clinical judgment.

i) Acute symptoms must have resolved and there are no sequelae that would place the participant at a higher risk of receiving study intervention, based on investigator Assessment. No repeat/follow-up COVID-19 testing is required

11 Subject has any condition that confounds the ability to interpret data from the study.

12 Subject has any of the following laboratory abnormalities: A. Absolute neutrophil count (ANC) < 1,000/µL. It is not permissible to administer GCSF to achieve minimum ANC levels within 7 days prior to screening complete blood count (CBC) (or within 14 days prior for pegfilgrastim).* B. Platelet count: < 75,000/µL for subjects in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count < 50,000/µL for subjects in whom ≥ 50% of bone marrow nucleated cells are plasma cells (transfusions are not permitted within 7 days prior to screening CBC).* C. Hemoglobin < 8 g/dL (< 4.9 mmol/L).*

* Participants who do not meet criteria for hematologic function because of MM-related cytopenias (e.g. due to extensive marrow involvement by MM) may receive transfusions and be screened after 1 week of transfusion.

D. Estimated glomerular filtration rate (eGFR) < 30 mL/min or requiring dialysis. eGFR will be calculated using the Modification of Diet in Renal Disease (MDRD) formula.

E. Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L) F. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × upper limit of normal (ULN) G. Serum total bilirubin > 1.5 × ULN, or for participants with documented Gilbert's syndrome > 3.0 mg/dL 13 Subject has peripheral neuropathy ≥ Grade 2 14 Subject with gastrointestinal disease or surgery (e.g., gastric bypass surgery) that may significantly alter the absorption of mezigdomide and/or other oral study treatment.

A. Subject has a prior history of malignancies other than MM, except if the participant has been free of the disease for ≥ 3 years. Patients with CIS treated with curative intent are not excluded if less than 3 years. Exceptions would include basal cell and squamous cell cancer of the skin treated with curative intent.

15 Subject has received immunosuppressive medication within the last 14 days of initiating study treatment. The following are exceptions to this criterion: a. Intranasal, inhaled, topical or local corticosteroid injections (e.g., intra-articular injection). b. Systemic corticosteroids at doses that do not exceed 10 mg/day of prednisone or the equivalent. c. Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication).

16 Administration of strong CYP3A modulators; administration of proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, pantoprazole, rabeprazole) within 2 weeks of starting study treatment.

17 Impaired cardiovascular function or clinically significant cardiovascular diseases, defined as any of the following within 6 months prior to enrollment: A. Acute myocardial infarction or acute coronary syndromes (eg, unstable angina, coronary artery bypass graft, coronary angioplasty or stenting, symptomatic pericardial effusion); B. Clinically significant cardiac arrhythmias (eg, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia); C. Thromboembolic or cerebrovascular events (eg, transient ischemic attack, cerebrovascular accident, deep vein thrombosis [unless associated with a central venous access complication] or pulmonary embolism); D. Prolonged QT syndrome (or QTcF > 470 msec at screening); E. LVEF <40% as determined by a MUGA scan or echocardiography. 18 Subject has uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment.

19 Subject who has had a live vaccine within 3 months of start of study therapy.

20 Subject is unable or unwilling to undergo protocol required thromboembolism or antiviral prophylaxis.

21 Subject is positive for human immunodeficiency virus (HIV), chronic or active hepatitis B, active hepatitis A, or active hepatitis C: A. Known positive HIV status. B. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg] either acute or chronic hepatitis). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBcAb] and/or antibodies to hepatitis B surface antigen [anti-HBsAb]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded.

EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.

EXCEPTION: Subjects with positive anti-HBcAb but negative HBsAg and negative anti-HBsAb profiles are eligible if HBV DNA PCR is negative.

C. Known to be seropositive for hepatitis C virus (HCV); anti-HCV antibody positive and HCV- ribonucleic acid (RNA) quantitation positive.

22 Subject has a history of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, pomalidomide (including ≥ Grade 3 rash during prior IMiD therapy), or dexamethasone or the excipients contained in the formulations, or subject has any contraindications per local PI.

23 Ongoing Grade 3 or higher peripheral sensory or motor neuropathy, history of Guillan-Barre syndrome (GBS) or GBS variants, or history of any Grade > 3 peripheral motor polyneuropathy.

24 Subject is an individual who is pregnant, nursing or breastfeeding, or who intends to become pregnant during participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From C1D1 to confirmed PD, lost to follow-up, or death (whichever occurs first), assessed up to 24 months
  Percentage of subjects who achieve best response of partial response (PR) or better according to the IMWG Uniform Response Criteria for Multiple Myeloma

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From randomization to first documentation of progressive disease or death due to any cause, assessed up to 24 months.
  Time from randomization to first documentation of progressive disease (PD) according to the IMWG Uniform Response Criteria for Multiple Myeloma (Kumar, 2016) or death due to any cause, whichever occurs first.
Overall survival (OS) | Time from randomization to time of death due to any cause, assessed up to 24 months.
Complete Response Rate (CR) or better | From C1D1 to confirmed PD, lost to follow-up, or death (whichever occurs first), assessed up to 24 months
  Percentage of subjects who achieve best response of complete response (CR) or better according to the IMWG Uniform Response Criteria for Multiple Myeloma (Kumar, 2016).
Very Good Partial Response Rate (VGPR) or better | From C1D1 to confirmed PD, lost to follow-up, or death (whichever occurs first), assessed up to 24 months
  Percentage of subjects who achieve best response of very good partial response (VGPR) or better according to the IMWG Uniform Response Criteria for Multiple Myeloma (Kumar, 2016).
Time to Response (TTR) | Time from randomization to the first documentation of response (PR or better), assessed up to 24 months.
Duration of Response (DOR) | Time from the first documentation of response (PR or better) to the first documentation of PD or death due to any cause, whichever occurs first, assessed up to 24 months.
Recommended mezigdomide dose | through study part 1 completion, up to 6 weeks.
  Recommended mezigdomide dose for Part 2, based on the totality of safety, and efficacy
Time to Next Treatment (TTNT) | Time from randomization to the start of the next antimyeloma treatment, assessed up to 24 months.
Safety profile (Adverse event) | From C1D1 to End of trial, assessed up to 24 months.
  Type, frequency, seriousness and severity of adverse events (AEs), and relationship of AEs to study treatment This includes frequency of grade 3/4 cytopenias and infection.
Minimal Residual Disease (MRD) negativity rate | From C1D1 to confirmed PD, lost to follow-up, or death (whichever occurs first), assessed up to 24 months
  Proportion of subjects who achieve complete response (CR) or better and are MRD negative

OTHER OUTCOMES:
Biomarkers | From C1D1 to End of trial, assessed up to 24 months.
  Correlation of baseline RNA/protein expression, gene expression, cytogenetics, copy number abnormalities and/or mutations in tumor cells to treatment response.
  Correlation of changes in RNA/protein expression, gene expression or genomic abnormalities in tumor cells to disease progression

CONTACTS AND LOCATIONS:
Locations (7):
- Singapore (2):
  - National University Hospital (NUH), Singapore
  - Singhealth Duke NUS blood cancer center, Singapore
- South Korea (5):
  - Chonnam National University Hwasun Hospital, Hwasun
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Seoul

IPD SHARING:
Plan to Share IPD: Undecided